CLINICAL TRIAL: NCT03305068
Title: Evaluation of Post-Procedure Administration of Celecoxib Following Shoulder Surgery: A Randomized Controlled Study
Brief Title: Evaluation of Post-Procedure Administration of Celecoxib Following Shoulder Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Louis Joint Replacement Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: BI177194
Record Dates: First submitted 2014-02-07; First posted 2017-10-09 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Reverse or Primary Total Shoulder; Rotator Cuff- Full Thickness- Repair
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- the use of a COX-II inhibitor in shoulder surgery. (Placebo Comparator): Arm 1 shoulder replacement, both primary and reverse
  Interventions: Drug: Celecoxib
- the use of a COX-II inhibitor in arhroscopic shoulder surgery. (Placebo Comparator): Arm 2 arthroscopic rotator cuff repair
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
Hypothesis It is expected that shoulder surgery patients treated with celecoxib (Celebrex) will experience significantly reduced narcotic use as measured by pill count compared with controls at three and six weeks postoperatively.

Study Overview The proposed study will determine if there is benefit to the use of a COX-II inhibitor in shoulder surgery. This study will have two arms: Arm 1 (shoulder replacement, both primary and reverse) and Arm 2 (arthroscopic rotator cuff repair). These distinct arms are necessary because each surgery is distinct in terms of type of procedure, indications, and patient population. The patients in Arm 1 will undergo stratified randomization according to the type of arthroplasty (primary or reverse) to ensure a balanced representation of these patients within subgroups. All patients undergoing primary total shoulder replacement, reverse shoulder replacement, or arthroscopic rotator cuff repair will be eligible to participate in the appropriate arm of the study. Revision surgery patients will be excluded from both arms of the study. A maximum of 78 arthroscopic cuff repair patients, and 78 arthroplasty patients will be enrolled in each arm of the study. Baseline information will be obtained on each patient including baseline VAS for pain, baseline shoulder scores as outlined below, and baseline narcotic and anti-inflammatory medication use, if any. Patients will be randomized to receive celecoxib (Celebrex) 400 mg one hour prior to surgery or placebo; they will then continue to receive the same medication daily for 3 weeks postoperatively: celecoxib 200 mg twice daily or a placebo control. The primary outcome measure will be narcotic utilization as measured by narcotic pill count. Secondary outcome measures will include subjective measure of pain as measured by the VAS for pain, range of motion as measured by active forward elevation (at 6 weeks postoperatively) and three patient assessment scores: the Simple Shoulder Test (SST), the UCLA score, and the American Shoulder and Elbow Society score (ASES). Data will be obtained at follow-up visits three and six weeks postoperatively.

DETAILED DESCRIPTION:
Hypothesis It is expected that shoulder surgery patients treated with celecoxib (Celebrex) will experience significantly reduced narcotic use as measured by pill count compared with controls at three and six weeks postoperatively.

Study Overview The proposed study will determine if there is benefit to the use of a COX-II inhibitor in shoulder surgery. This study will have two arms: Arm 1 (shoulder replacement, both primary and reverse) and Arm 2 (arthroscopic rotator cuff repair). These distinct arms are necessary because each surgery is distinct in terms of type of procedure, indications, and patient population. The patients in Arm 1 will undergo stratified randomization according to the type of arthroplasty (primary or reverse) to ensure a balanced representation of these patients within subgroups. All patients undergoing primary total shoulder replacement, reverse shoulder replacement, or arthroscopic rotator cuff repair will be eligible to participate in the appropriate arm of the study. Revision surgery patients will be excluded from both arms of the study. A maximum of 78 arthroscopic cuff repair patients, and 78 arthroplasty patients will be enrolled in each arm of the study. Baseline information will be obtained on each patient including baseline VAS for pain, baseline shoulder scores as outlined below, and baseline narcotic and anti-inflammatory medication use, if any. Patients will be randomized to receive celecoxib (Celebrex) 400 mg one hour prior to surgery or placebo; they will then continue to receive the same medication daily for 3 weeks postoperatively: celecoxib 200 mg twice daily or a placebo control. The primary outcome measure will be narcotic utilization as measured by narcotic pill count. Secondary outcome measures will include subjective measure of pain as measured by the VAS for pain, range of motion as measured by active forward elevation (at 6 weeks postoperatively) and three patient assessment scores: the Simple Shoulder Test (SST), the UCLA score, and the American Shoulder and Elbow Society score (ASES). Data will be obtained at follow-up visits three and six weeks postoperatively.

ELIGIBILITY:
Inclusion / Exclusion Criteria for Pfizer Study

Inclusion Criteria:

1. community ambulators
2. D/C to home only
3. only MO and IL pts
4. Primary unilateral shoulder replacements / Cuff tear
5. Full Thickness, single tendon tear

Exclusion Criteria:

1. allergy, sensitivity, or inability to take Celebrex
2. CR >1.5
3. h/o bleeding ulcers
4. h/o Inflammatory bowel disease, Crohn's disease, ulcerative colitis
5. Coagulation abnormality
6. Coumadin/Plavix/Xaralto
7. CHF
8. Previous MI or CVA
9. Current use of long acting narcotics (Fentanyl Patches, Oxycontin CR, MS Contin)
10. Refusal by PCP or cardiologist

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
This study will determine if use of celecoxib (Celebrex) for three weeks after shoulder surgery will reduce pain as measured by decreased narcotic consumption. | 3 weeks
This study will determine if use of celecoxib (Celebrex) for three weeks after shoulder surgery will reduce pain as measured by decreased narcotic consumption. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Burns, MD, Principal Investigator — SSM orthopedics
Locations (1):
- SSM DePaul, Bridgeton, Missouri, United States